CLINICAL TRIAL: NCT00237796
Title: Functional Rehabilitation of Older Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O3341-R
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-03

CONDITIONS: Psychotic Disorders; Schizoaffective Disorder; Schizophrenia
Keywords: Behavioral; Cognitive; Functioning; Older; CBT; Rehabilitation; Schizophrenia; Skills; Social; Training
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 1 (Experimental): Cognitive Behavioral Social Skills Training (CBSST)
  Interventions: Behavioral: Cognitive Behavioral Social Skills Training (CBSST)
- ARM 2 (Active Comparator): Goal Focused Supportive Contact (GFSC)
  Interventions: Behavioral: Goal Focused Supportive Contact (GFSC)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Social Skills Training (CBSST) — Thought challenging, social communication skills, and problem solving skills are trained in group therapy 2 hours per week for 9 months.
  Arms: ARM 1
Behavioral: Goal Focused Supportive Contact (GFSC) — Active goal setting and supportive contact in group therapy 2 hours per week for 9 months.
  Arms: ARM 2

SUMMARY:
The primary purpose of this project is to evaluate the efficacy of a group therapy intervention, cognitive behavioral social skills training (CBSST), that teaches social functioning skills and cognitive-behavioral compensatory aids to older patients with schizophrenia. CBSST, therefore, targets the multidimensional deficits that lead to disability in aging veterans with severe mental illness.

DETAILED DESCRIPTION:
This is a randomized-controlled clinical trial comparing 2 treatment conditions: Goal focused supportive care (SC); and CBSST. Subjects (N=100) will be recruited, treated for 9 months and followed longitudinally for 9 months after treatment. A multidimensional evaluation of treatment outcome, including social functioning (primary outcome), neuropsychological functioning, cognitive insight, psychotic symptoms, and health services utilization, will be conducted at baseline, end of treatment (9-month follow-up), and 9 months post-treatment. 100 patients with schizophrenia or schizoaffective disorder will participate on a voluntary basis and will be paid $50.00 per assessment visit. Subjects will not be paid or given any incentive for treatment. The following inclusion/exclusion criteria will be used: (i) Voluntary informed consent for participation (given by the patient or conservator); (ii) Age 45 or older; (iii) DSM-IV-diagnosis (APA, 1994) of schizophrenia or schizoaffective disorder at any stage of illness; (iv) No prior exposure to SST or CBT in the past 5 years; (v) Level of care required at baseline does not interfere with outpatient group therapy participation (e.g., partial or inpatient hospitalization for psychiatric, or physical illness). We anticipate that we will be able to provide an empirically validated intervention that can be used by clinicians on multidisciplinary rehabilitation teams to reduce disability in aging patients with schizophrenia. The products from this research will be written research reports and a therapy manual and patient workbook to guide rehabilitation that can be disseminated (e.g., via the internet) to relevant clinicians.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age and older
* DSM-IV diagnosis of Schizophrenia or Schizoaffective Disorder
* Fluent in speaking, reading, and writing English
* Physically and psychiatrically stable enough to undergo various assessments in this study

Exclusion Criteria:

Has not received Cognitive Behavioral Therapy (CBT) or Social Skills Training (SST) or Dialectical Behavioral Therapy (DBT) in the past 5 years

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Granholm, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Result] Granholm E, Holden J, Link PC, McQuaid JR, Jeste DV. Randomized controlled trial of cognitive behavioral social skills training for older consumers with schizophrenia: defeatist performance attitudes and functional outcome. Am J Geriatr Psychiatry. 2013 Mar;21(3):251-62. doi: 10.1016/j.jagp.2012.10.014. Epub 2013 Jan 10. PMID 23395192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included 79 middle age and older community dwelling Veteran and non-veterans. Inclusion criteria: diagnosis of schizophrenia or schizoaffective, age 45 or older, and fluency in English. Exclusion criteria: prior exposure to CBT during the previous five years.
Pre-assignment Details: Baseline data were collected before randomization. N=116 participants enrolled in the study and N=79 started.
  Total of 37 excluded for reasons: n=20 lost interest; n=6 wrong diagnosis, n=3 not psychiatrically stable; n=3 not medically stable, and n=5 lost contact/moved.
Groups:
- Cognitive Behavioral Social Skills Training (CBSST): Cognitive Behavioral Social Skills Training: Thought challenging, social communication skills, and problem solving skills are trained in group therapy 2 hours per week for 9 months.
- Goal Focused Supportive Contact (GFSC): Goal Focused Supportive Contact: Active goal setting and supportive contact in group therapy 2 hours per week for 9 months.
Period: Overall Study
Arm/Group | Cognitive Behavioral Social Skills Training (CBSST) | Goal Focused Supportive Contact (GFSC)
Started | 41 | 38
Completed | 31 | 33
Not Completed | 10 | 5
Not completed — Baseline and one other ILSS required | 10 | 5

BASELINE CHARACTERISTICS:
Population: Participants numbers reported include at least one baseline and at least 1 ILSS assesssment
Groups:
- Goal Focused Supportive Contact (GFSC): Goal Directed Supportive Care Contact: Active goal setting and supportive contact in group therapy 2 hours per week for 9 months.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Social Skills Training (CBSST) | Goal Focused Supportive Contact (GFSC) | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Customized [Number; unit: participants]
  Between ages 45 to 78 | 31 | 33 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Independent Living Skills Survey (ILSS)
Description: The ILSS is a self-report measure in an interview format to assess everyday functioning in ten domains: Appearance and Clothing, Personal Hygiene, Care of Personal Possessions, Food Preparation/Storage, Health Maintenance, Money Management, Transportation, Leisure, Job Seeking, and Job Maintenance. Scale ranges from 0 to 1. Subscales are averaged to yield composite score. Higher scores represent higher level of functioning.
Time Frame: baseline, mid-treatment, end of treatment, mid-follow up, and follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Social Skills Training: Cognitive Behavioral Social Skills Training: Thought challenging, social communication skills, and problem solving skills are trained in group therapy 2 hours per week for 9 months.
- Goal Focused Supportive Contact: Goal Focused Supportive Contact
  Goal Focused Supportive Contact: Active goal setting and supportive contact in group therapy 2 hours per week for 9 months.
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 0.66 (0.09) | 0.70 (0.11)
  Mid-treatment (4.5 months) | 0.68 (0.10) | 0.71 (0.10)
  End of treatment (9 months) | 0.68 (0.07) | 0.71 (0.12)
  Mid-Followup (13.5 months) | 0.68 (0.07) | 0.72 (0.12)
  Follow Up (9 months) | 0.71 (0.07) | 0.68 (0.13)

2. Secondary Outcome: Comprehensive Module Test (CMT)
Description: The Comprehensive Module Test (CMT) is an assessment of CBSST skills acquisition in three domains: Communication Skills Test, Problem Solving Test, and Thought Challenging Test. The total CMT score ranges from 0-33. Higher total scores represent higher level of CBSST skills acquisition.
Time Frame: baseline, mid-treatment, end of treatment, mid-follow up, and follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Goal Focused Supportive Contact: Goal Focused Supportive Contact: Active goal setting and supportive contact in group therapy 2 hours per week for 9 months.
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 6.2 (3.6) | 4.8 (3.3)
  Mid-treatment (4.5 months) | 8.6 (5.6) | 6.2 (5.1)
  End of treatment (9 months) | 12.0 (7.1) | 5.5 (4.1)
  Mid-Followup (13.5 months) | 10.5 (4.8) | 6.3 (4.3)
  Follow Up (9 months) | 11.2 (7.2) | 5.8 (3.8)

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) - Positive Subscale
Description: The PANSS is 30 item semi-structured clinical interview designed to assess positive and negative symptoms. Positive symptoms are rated on 7 domains: Delusions, Conceptual Disorganization, Hallucinatory Behavior, Excitement, Grandiosity, Suspiciousness/Persecution, and Hostility. Each domain in the positive symptom subscale is rated from 0 (absence of symptom) to 7 (extreme symptom severity). Total scores of the seven domains are summed to yield a total score range of 0 (Absence) to 49 (Extreme), where higher scores represent more severe positive symptoms.
Time Frame: baseline, mid-treatment, end of treatment, mid follow-up, and followup
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 18.3 (8.1) | 17.8 (6.3)
  Mid-treatment (4.5 months) | 17.4 (6.4) | 15.5 (5.8)
  End of treatment (9 months) | 15.5 (5.8) | 16.1 (5.3)
  Mid-Followup (13.5 months) | 15.8 (6.8) | 18.0 (6.7)
  Follow Up (9 months) | 15.7 (5.5) | 18.5 (8.1)

4. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS) - Diminished Expression
Description: The SANS is a 25 item semi-structured clinical interview designed to assess negative symptoms. The first 13 items measure diminished expression which consists of two domains: Affective flattening and Alogia. Each item is rated from 0 (Absent) to 5 (Severe). The total score is derived from the average of the Affective Flattening and Alogia global ratings (items #8 and #13).
Time Frame: baseline, mid treatment, end of treatment, mid follow-up, and follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 1.63 (1.37) | 1.79 (1.09)
  Mid-treatment (4.5 months) | 1.72 (1.13) | 1.48 (0.87)
  End of treatment (9 months) | 1.21 (1.12) | 1.38 (1.04)
  Mid-Followup (13.5 months) | 1.71 (1.00) | 1.62 (1.31)
  Follow Up (9 months) | 1.62 (1.06) | 1.83 (1.30)

5. Secondary Outcome: The Scale for the Assessment of Negative Symptoms (SANS) - Diminished Motivation
Description: The SANS is a 25 item semi-structured clinical interview designed to assess negative symptoms. There are 9 items that measure diminished motivation which consists of two domains: Avolition-Apathy and Anhedonia-Asociality. Each item is rated from 0 (Absent) to 5 (Severe). The total score is derived from the average of the Affective Flattening and Alogia global ratings (items #17 and #22).
Time Frame: baseline, mid-treatment, end of treatment, mid follow-up, and follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 2.02 (1.17) | 2.46 (1.15)
  Mid-treatment (4.5 months) | 2.09 (1.35) | 2.15 (1.18)
  End of treatment (9 months) | 1.90 (1.30) | 1.83 (1.31)
  Mid-Followup (13.5 months) | 1.53 (1.03) | 1.92 (1.43)
  Follow Up (9 months) | 1.72 (1.02) | 1.93 (1.44)

6. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a self-report measure of depression that consists of 21 questions. The total scale ranges from 0-63. Scores from individual questions are summed to yield a total score. Higher scores represent greater severity of depression.
Time Frame: baseline, mid-treatment, end of treatment, mid follow-up, and follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 16.3 (9.8) | 16.4 (13.5)
  Mid-treatment (4.5 months) | 17.2 (12.3) | 13.8 (11.2)
  End of treatment (9 months) | 15.0 (12.6) | 14.3 (14.0)
  Mid-Followup (13.5 months) | 9.1 (7.9) | 12.9 (12.7)

7. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The Beck Anxiety Inventory is a self-report measure of anxiety that consists of 21 questions. Scores from individual items are summed to yield a total score. The total score ranges from 0-63. Higher scores represent greater severity of anxiety.
Time Frame: baseline, mid-treatment, end of treatment, mid follow-up, and follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Skills Training | Goal Focused Supportive Contact
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 16.4 (12.7) | 14.5 (12.1)
  Mid-treatment (4.5 months) | 14.2 (12.3) | 12.4 (12.1)
  End of treatment (9 months) | 15.7 (14.2) | 10.6 (10.1)
  Mid-Followup (13.5 months) | 12.3 (12.2) | 10.5 (11.4)
  Follow Up (9 months) | 11.5 (10.1) | 10.4 (11.0)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- CBSST: Cognitive Behavioral Social Skills Training: Thought challenging, social communication skills, and problem solving skills are trained in group therapy 2 hours per week for 9 months.
- Goal Directed Supportive Care: Goal Directed Supportive Care Contact: Active goal setting and supportive contact in group therapy 2 hours per week for 9 months.
Arm/Group | CBSST | Goal Directed Supportive Care
Serious Adverse Events (participants affected / at risk) | 4/41 | 11/38
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBSST (N=41) | Goal Directed Supportive Care (N=38)
Hospitalization (Psychiatric disorders) | 2 (4) | 9 (18)
Hospitalization (Endocrine disorders) | 1 (1) | 0 (0)
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
* Randomization of treatment groups were not matched on the primary outcome (ILSS) at baseline but this was controlled using baseline ILSS as a covariate.
* Participant dropout varied across assessments

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No